CLINICAL TRIAL: NCT05317923
Title: Airway Management During Unusual Tracheal Stenosis: A Clinical Feasibility Trial
Brief Title: Airway Management During Unusual Tracheal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, Associate Professor, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/1958
Record Dates: First submitted 2022-03-14; First posted 2022-04-08 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Tracheal Stenosis
Keywords: prolonged intubation,; tracheal stenosis; Covid-19
MeSH Terms: conditions — Tracheal Stenosis; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- airway management and ventilation in patients with unusual placement of tracheal stenosis (Experimental): Flow-controlled ventilation (FCV) in patients with unusual placement of tracheal stenosis
  Interventions: Other: Flow Controlled Ventilation

INTERVENTIONS:
Other: Flow Controlled Ventilation — Anesthesia management in patients with subglottic tracheal stenosis with flow-controlled ventilation using an intubation tube with an inner diameter of less than 3 mm

SUMMARY:
Tracheal stenosis is a serious complication following prolonged intubation. There are important differences in the challenges of airway management. This study consists of our anesthesia management experience in patients with unusual placement of tracheal stenosis due to Covid-19 undergoing tracheal dilatation.

DETAILED DESCRIPTION:
Tracheal stenosis is a serious complication following prolonged intubation. Two types of tracheal stenosis; Glottic and subglottic stenoses have common features in that they are challenging in terms of ventilation, oxygenation and intubation. However, there are important differences in the challenges of airway managementA thinner tube may be sufficient to overcome the airway difficulty in glottic stenoses. However, in subglottic tracheal stenosis, a thinner tube may not be conveyed to the distal of the stenosis. As a result, adequate ventilation and oxygenation may not be provided with an intubation tube placed proximal to the trachea. This study consists of our anesthesia management experience in patients with unusual placement of tracheal stenosis due to Covid-19 undergoing tracheal dilatation.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3 patients over the age of 18 who are scheduled for an elective laryngeal procedure due to subglottic stenosis will be included in our study.

Exclusion Criteria:

1. Patients who did not agree to participate in the study.
2. Congestive heart failure (ejection fraction ≤ 35 %)
3. Emergency laryngeal procedures.
4. Patients under 18 years old.
5. Patients with ASA > 3.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
PCO2 | PCO2 value at baseline just before entubation, peroperative 5, 15, 30, 45 minutes after induction, and before the extubation through surgery completion
  blood partial pressure of carbondioxide
PO2 | PO2 value at baseline just before entubation, peroperative 5, 15, 30, 45 minutes after induction, and before the extubation through surgery completion
  blood partial pressure of oxygen

SECONDARY OUTCOMES:
EtCO2 | EtCO2 value at baseline just before entubation, peroperative 5, 15, 30, 45 minutes after induction, and before the extubation through surgery completion
  end-tidal carbondioxide measurement
length of intubation due to Covid-19 Pnomonia | postoperative period (up to 1 year)
  time from intubation to extubation in ICU
sPO2 | SPO2 value at baseline, peroperative 5, 15, 30, 45 minutes after induction, and before the extubation through surgery completion
  peripheral oxygen saturation
Myers-Cotton grading scale (1/2/3) | before the surgery
  The grade of tracheal stenosis
VAS (Visual Analogue Scale) score (between 0 to 10 points) | during surgery through surgery completion
  surgeons' satisfaction(VAS 0=the worst view, 10= the best view)

CONTACTS AND LOCATIONS:
Overall Officials: Istnabul University, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No